CLINICAL TRIAL: NCT00966498
Title: Peripheral Blood Stem Cell Transplantation in Children With High-Risk or Recurrent Solid Tumors
Brief Title: Peripheral Blood Stem Cell Transplant (PBSCT) in Children With High Risk or Recurrent Solid Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kuang-Yueh Chiang, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1023-2003; PBSCT for ST (Other: Other)
Record Dates: First submitted 2009-08-11; First posted 2009-08-27 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: High Risk Solid Tumors; Recurrent Solid Tumors
Keywords: malignancy; solid tumor; recurrent; high risk
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): This study is a single-arm, non-randomized trial. Peripheral blood stem cells will be harvested by mobilization with chemotherapy followed by G-CSF. Following adequate peripheral blood stem cell collection, the patients would be transplanted using the conditioning regimen consisting of thiotepa and cyclophosphamide (tandem one) and busulfan and melphalan (tandem two). They will receive G-CSF post transplant. There will be 6-8 weeks interval between tandem transplants. All patients would be carefully observed for any toxicity, transplant-related complications, relapse and disease-free survival.
  Interventions: Procedure: Peripheral Blood Stem Cell Transplant

INTERVENTIONS:
Procedure: Peripheral Blood Stem Cell Transplant — Peripheral Blood Stem Cell Transplant

SUMMARY:
Before the transplant, the patient will have a pre-transplant evaluation. This will help find out whether there are health problems that will prevent the transplant. It also provides "baseline" tests that will be used later to see whether or not organs have gotten better or worse after the transplant. Prior to the stem cell collection, the patient will get chemotherapy to help try to put him/her in remission and to push more stem cells into the peripheral blood (mobilization). The study doctor will decide which chemotherapy will be used for this part of the study. Once mobilization is completed, the peripheral blood stem cell collection (apheresis) will be done in the clinic. The apheresis machine will draw blood out of the central line. The blood then passes through the apheresis machine and the stem cells are separated out. The remaining blood is sent back through the central line. If the investigators are unable to collect enough peripheral blood stem cells, a bone marrow harvest may be necessary to collect more stem cells.

The patient will then be admitted to the hospital for the first transplant. He/she will get Thiotepa and Cyclophosphamide. Then the patient will be given back the cells that were collected. The cells are given in the same manner as a blood transfusion. The patient will be kept in the hospital until he/she is stable and blood counts are increasing. Approximately 6 to 8 weeks after Day 0 of the 1st transplant, the patient will be admitted for the second transplant. At this time, he/she will get Busulfan and Melphalan and then the collected cells will be given back. The patient will be kept in the hospital until he/she is stable and blood counts are increasing. Frequent clinic follow-up is required.

This study is open to patients who are less then 21 years of age with refractory or relapsed high-risk, solid tumors, excluding neuroblastoma (there is a cooperative group trial for these patients). Patients will be identified by the Transplant team and eligibility will be verified by a member of the clinical research team. Patients will be cared for by members of the Transplant team and various other subspecialty physicians.

DETAILED DESCRIPTION:
The optimal treatment for refractory (disease won't go away with standard treatment) or relapsed (disease comes back after going away) solid tumors is unknown. Recent studies have shown some benefit to tandem peripheral blood stem cell transplantation (PBSCT). In a tandem transplant, two transplants are done, one after the other. To do a PBSCT, stem cells ("mother cells" that can become any other type of cell) are first collected from the patient's circulating blood. The patient then undergoes high-dose chemotherapy called the preparative regimen. The preparative regimen destroys not only the tumor cells, but it also destroys all of the normal blood making cells. The collected cells are then given back to the patient to "rescue" the patient from the devastating effects of the preparative regimen. By using a stem cell rescue will are able to give much higher doses of chemotherapy than we would be able to give without the stem cell rescue. To make sure that all of the tumor cells are destroyed, patients in this study will undergo two separate transplants using two different preparative regimens. The preparative regimens will use the best agents that have been found to work against recurrent and refractory solid tumors: Busulfan, Thiotepa, Cyclophosphamide and Melphalan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with high risk recurrent or refractory solid tumors following initial chemotherapy
2. Tumor must be sensitive to chemotherapy (maximum 8 cycles) and/or radiation defined as a greater than 50% reduction in size of the primary and/or metastatic sites.
3. Patients who are under 35 years of age.
4. Patients with a life expectancy of at least 8 weeks and performance status (Karnofsky or Lansky score) of at least 70%.
5. Patients who are acceptable candidates for peripheral blood stem cell transplantation based on their pre-transplant evaluation.

Exclusion Criteria:

1. Patients will not be excluded based on sex, race.
2. Patients with central nervous system tumors are not eligible for this protocol.
3. Patients have significant functional deficits in major organs which would interfere with successful outcome following PBSCT.
4. Patients who have been treated for infections must have appropriate responses as documented by negative cultures and/or a normal radiographic examination.
5. Patients may not have active CNS disease or marrow involvement with the tumor at the time of transplant.
6. Patients with disease progression after tandem PBSC #1 will not be eligible for tandem PBSC #2.
7. Patients will be excluded if they are women of childbearing potential who are currently pregnant (HCG+) or who are not practicing adequate contraception.
8. Patients who have had a previous stem cell transplant.

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2003-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility and toxicity of tandem high dose chemotherapy and peripheral blood stem cells rescue in patients with high-risk or recurrent solid tumors. | 1 year after last patient is enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Yueh Chiang, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia